CLINICAL TRIAL: NCT00366951
Title: A Randomized Clinical Trial Comparing the Efficacy and Safety of Foley Catheter Balloon With Oxytocin and Extraamniotic Saline Infusion (EASI) With Oxytocin for Induction of Labor Requiring Cervical Ripening
Brief Title: A Randomized Study on Comparing the Efficacy of Foley Catheter and Extraamniotic Saline Infusion for Labor Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ORA#: 03111102
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Cervical Ripening; Labor, Induced
Keywords: Cervical Ripening; Labor, Induced; Balloon Dilation; Oxytocin

INTERVENTIONS:
Procedure: Foley catheter only
Procedure: Extraamniotic saline infusion

SUMMARY:
Our purpose was to compare the efficacy and safety of Foley catheter with oxytocin and extraamniotic saline infusion with oxytocin for induction of labor requiring cervical ripening.

DETAILED DESCRIPTION:
Induction of labor is indicated when the benefit to either the mother or fetus outweighs that of continuing the pregnancy. Labor induction in the presence of an unripened cervix is associated with prolonged labor, chorioamnionitis, and cesarean delivery. Numerous mechanical and pharmacological methods have been used for cervical ripening. There are limited numbers of rigorous studies comparing the efficacy of the various methods. One of the most common mechanical methods for cervical ripening is placement of a Foley catheter with a 30 cc balloon inside the cervix, with or without the use of oxytocin. The Foley balloon will disrupt the amniotic membrane surface and cause the release of prostaglandin, a natural chemical from the cervix, to facilitate the ripening process. Oxytocin will be used concurrently as the induction agent. Recently, a modification of this method, extraamniotic saline infusion (EASI) has become more popular. The EASI method involves similar procedure including the placement of Foley catheter inside the cervix; in addition, saline solution will be infused through the catheter. This additional step is thought to further facilitate the disruption of amniotic membrane surface. Both methods are safe and become the standard treatment for cervical ripening. However, there are no published trials so far comparing the two methods. The objective of this study is to compare the efficacy and safety of Foley catheter with oxytocin and EASI with oxytocin for induction of labor requiring cervical ripening. The study is designed to be a single masked randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* singleton gestation
* cephalic vertex presentation
* intact membrane
* gestational age between 30 and 42 weeks
* Bishop score less than or equal to 5

Exclusion Criteria:

* suspected chorioamnionitis
* placenta previa
* low lying placenta
* unexplained vaginal bleeding
* intrauterine fetal demise
* HIV
* any contraindication to vaginal delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2004-04; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The time interval from placement of Foley catheter to vaginal delivery

SECONDARY OUTCOMES:
Cesarean delivery rate
Incidence of maternal complications
Incidence of neonatal complications

CONTACTS AND LOCATIONS:
Overall Officials: Yukmei R Lam, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264